CLINICAL TRIAL: NCT01530646
Title: Molecular Events Underpinning Changes in Tissue Metabolism With Whey and Soy Ingestion in Energy Restriction in Overweight/Obese Adults
Brief Title: Impact of Whey and Soy Protein Ingestion in Conjunction With Energy Restriction in Overweight/Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart M. Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-999
Record Dates: First submitted 2011-08-04; First posted 2012-02-10 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
Keywords: obesity; overweight; muscle; protein; muscle protein synthesis; muscle protein breakdown; whey; soy; caloric restriction
MeSH Terms: conditions — Obesity; Overweight | interventions — Whey

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator): Carbohydrate & 750 kcal dietary restriction while they receive a daily supplement (2 x 25 g) of maltodextrin (no protein) for 14 days. Weight loss.
  Interventions: Behavioral: Weight loss
- Whey (Experimental): Whey protein & 750 kcal dietary restriction while they receive a daily supplement (2 x 25 g) of WPI for 14 days. Weight loss.
  Interventions: Behavioral: Weight loss; Dietary Supplement: Whey
- Soy (Experimental): Soy protein & 750 kcal dietary restriction while they receive a daily supplement (2 x 25 g) of SPC for 14 days. Weight loss.
  Interventions: Behavioral: Weight loss; Dietary Supplement: Soy

INTERVENTIONS:
Behavioral: Weight loss — -750kcal/d
Dietary Supplement: Soy — 2 x 25g/d SPC
  Arms: Soy
Dietary Supplement: Whey — 2 x 25g/d WPI
  Arms: Whey

SUMMARY:
It is known that dieting (restricted energy intake) without resistance training leads to a reduced metabolic rate, and the loss of both fat and muscle mass. When exercise is not included in a period of restricted energy intake, the degree to which muscle mass is lost is highly dependent upon protein consumption. Whey protein is a high quality protein isolated from milk and is known to stimulate new protein synthesis for all proteins in your body. Previous research has established that the consumption of whey protein has been correlated with retaining muscle mass while stimulating fat loss. However, the mechanisms behind these findings is still unknown. The purpose of this study is to establish a mechanistic underpinning to the efficacy of whey protein versus soy protein and a carbohydrate control (maltodextrin), in promoting fat mass loss and lean mass retention during a period of short-term controlled dietary energy deficit (-750 kcalories/day).

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 to 55 years old
* Moderately Obese/Overweight (body mass index > 25 and < 42 kg/m2)
* Healthy
* Non-smoker

Exclusion Criteria:

* Suffer from type 2 diabetes, hyperlipidemia, or thyroid dysfunction
* Taking medications
* Having an unstable weight in the past 4-6 months, or dieting at some time during the past 6 months
* Taking weight loss products or aids (including energy drinks)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis rate and lipolytic rate as measured using stable isotope and glycerol infusions. | After 14 day dietary intervention

SECONDARY OUTCOMES:
Transcriptomic changes (via gene profiling) associated with the effects of whey on lipogenic and lipid oxidative genes, and protein synthetic pathways in muscle. | After 14 days of dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, Ph.D., Principal Investigator — Department of Kinesiology, McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Hector AJ, Marcotte GR, Churchward-Venne TA, Murphy CH, Breen L, von Allmen M, Baker SK, Phillips SM. Whey protein supplementation preserves postprandial myofibrillar protein synthesis during short-term energy restriction in overweight and obese adults. J Nutr. 2015 Feb;145(2):246-52. doi: 10.3945/jn.114.200832. Epub 2014 Dec 17. PMID 25644344
- [Derived] Paschalis V, Theodorou AA, Margaritelis NV, Kyparos A, Nikolaidis MG. N-acetylcysteine supplementation increases exercise performance and reduces oxidative stress only in individuals with low levels of glutathione. Free Radic Biol Med. 2018 Feb 1;115:288-297. doi: 10.1016/j.freeradbiomed.2017.12.007. Epub 2017 Dec 9. PMID 29233792
- [Derived] Churchward-Venne TA, Breen L, Di Donato DM, Hector AJ, Mitchell CJ, Moore DR, Stellingwerff T, Breuille D, Offord EA, Baker SK, Phillips SM. Leucine supplementation of a low-protein mixed macronutrient beverage enhances myofibrillar protein synthesis in young men: a double-blind, randomized trial. Am J Clin Nutr. 2014 Feb;99(2):276-86. doi: 10.3945/ajcn.113.068775. Epub 2013 Nov 27. PMID 24284442
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/25644344